CLINICAL TRIAL: NCT01800955
Title: The Effectiveness of Resistive Capacitive Diathermy in Patients Affected by Knee Osteoarthritis: a Sham-controlled Study
Brief Title: Effectiveness of Resistive Capacitive Diathermy in Patients Affected by Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Bertolini, Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1347/2012
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Knee Osteoarthritis
Keywords: physical therapy; diathermy; knee; osteoarthritis; pain; physical function
MeSH Terms: conditions — Osteoarthritis, Knee; Fever; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- resistive capacitive diathermy (Experimental): in the resistive capacitive diathermy protocol patients are administered the resistive capacitive diathermy treatment for a thirty minutes session, three times per week for a total of ten sessions
  Interventions: Device: resistive capacitive diathermy treatment (resistive capacitive diathermy, Hcr 902, Unibell)
- sham placebo group (Sham Comparator): The sham treatment is administered with the resistive capacitive diathermy device set on "on" but not active (not supplying energy) with the same type of application, the same frequency and duration of experimental diathermy group
  Interventions: Other: sham placebo resistive capacitive diathermy treatment

INTERVENTIONS:
Device: resistive capacitive diathermy treatment (resistive capacitive diathermy, Hcr 902, Unibell) — The resistive capacitive diathermy is a medical device supplying low (448 KHz) radiofrequencies with maximum output power of 200 W. It is used to reduce pain and inflammation and allowing healing processes. diathermy treatment is administered for a thirty minutes session, three times per week for a total of ten sessions.
  Arms: resistive capacitive diathermy
Other: sham placebo resistive capacitive diathermy treatment — The sham treatment is administered with the diathermy device set on "on" but not active (not supplying energy) and the treatment session has the same modalities, frequency and duration of experimental diathermy group
  Arms: sham placebo group

SUMMARY:
It is a double-blind randomized sham-controlled clinical trial to evaluate the effectiveness of resistive capacitive diathermy in subjects affected by knee osteoarthritis in comparison with a "sham" diathermy treatment. The resistive capacitive diathermy is a medical device supplying low (448 KHz) radiofrequencies with maximum output power of 200 W, used to reduce pain and inflammation and allowing healing processes. The sham diathermy treatment is administered with the device set on "on" but not active (not supplying energy). Each subject, randomly assigned to either resistive capacitive diathermy treatment (group 1) or sham-treatment (group 2) is submitted to a thirty minutes session, three times per week for a total of ten sessions. The outcome measures are the WOMAC scale (Western Ontario and McMaster Universities Arthritis Index) to assess pain and physical functioning, a visual analogic scale (VAS) for pain, the femoral quadriceps strength (MRC = Medical Research Council Scale). Outcome measures are administered at baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2) and 3 months (T3) after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Knee osteoarthritis established by clinical examination and X-ray in postero-anterior and lateral views

Exclusion Criteria:

* Neurologic Disorders involving the lower limbs
* Systemic inflammatory disorders
* pace-maker implantation
* Severe heart disease
* Acute infections or bone tuberculosis
* Acute skin diseases
* History of surgery on the affected knee
* Cognitive or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
changing of the Western Ontario and McMaster Universities Arthritis Index WOMAC)scale | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2) and 3 months (T3) after the end of treatment
  assessment of changing of pain and physical functioning in patients affected by osteoarthritis of lower limbs

SECONDARY OUTCOMES:
changing of visual analogic scale (VAS) | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2) and 3 months (T3) after the end of treatment
  assessment of changing of pain
MRC scale = Medical Research Council Scale | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2) and 3 months (T3) after the end of treatment
  assessment of changing of femoral quadriceps strength

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital "A. Gemelli", Catholic University of the Sacred Heart, Rome, Italy